CLINICAL TRIAL: NCT03385408
Title: Effectiveness of High-intensity Laser Therapy in Shoulder Osteoarthritis; a Prospective, Randomized, Controlled Study
Brief Title: Effectiveness of HILT in Shoulder Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Justyna Wyszyńska, Principal Investigator, University of Rzeszow
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HILT-osteoarthritis
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Osteoarthritis of the Shoulder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HILT group (Experimental): High-intensity laser therapy application through HIRO 3.0 device
  Interventions: Device: HIRO® 3.0
- Placebo group (Sham Comparator): Sham high-intensity laser therapy application through HIRO 3.0 device
  Interventions: Device: Sham laser

INTERVENTIONS:
Device: HIRO® 3.0 — Patients will receive pulsed Nd:YAG (yttrium aluminum garnet) laser, produced by HIRO 3.0 device (ASA, Vicenza, Italy). The total energy deliver to the patient during one session will be 3.000 J through three phases of treatment. HILT will be applied for a total of 4 weeks (three sessions/week).
  Arms: HILT group
Device: Sham laser — For sham laser, the patient will attended the physical therapy clinic three times a week for 4 weeks and receive sham laser. It is applies the same time than experimental one but with 0 W.
  Arms: Placebo group

SUMMARY:
This study will determine the efficacy of High Intensity Laser Therapy (HILT) for the treatment of shoulder osteoarthritis.

DETAILED DESCRIPTION:
Shoulder osteoarthritis (SO) is a musculoskeletal joint disease that affects the elderly. SO is characterized by degeneration of the articular cartilage in the involved joints and its underlying bone within a joint as well as bony overgrowth. It is one of the major causes of physical disability that has a social and public health impact due to pain, stiffness, joint instability, and muscle weakness.

The diagnosed patients with SO will be treated with HILT for a total of ten sessions during the entire duration of the treatment protocol. Parameters to be evaluated are: range of motion, pressure pain (algometer), pain perception (Visual Analog Scale (VAS), Modified Laitinen Pain Questionnaire), quality of life (WHOQoL-BREF) These parameters will be recorded before the first treatment (baseline), after completion of treatment, three and 12 months after completion treatment. A change in above parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. painful osteoarthritis of the shoulder for at least 6 months
2. not engage in any other treatment during treatment period
3. pain ≥4 on the visual analog scale (VAS) in the previous 3 months

Exclusion Criteria:

1. presence of any other musculoskeletal problems associated with the shoulder joint, such as fracture, tendon or ligament tears, meniscus injury, rheumatoid arthritis, or shoulder surgery
2. receiving physical therapy and/or intra-articular corticosteroid or hyaluronic acid injections during the last 6 months
3. absolute and relative contraindications of Laser Therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2019-08-21 (Actual)

PRIMARY OUTCOMES:
Change in the pain perception | at baseline, immediately after treatment completion, 3 and 12 months after treatment completion
  Evolution of pain (Visual Analogic Scale and the Modified Laitinen Pain Questionnaire) between baseline, after the end of the protocol treatment, 3 and 12 months after the end of the protocol treatment

SECONDARY OUTCOMES:
Change in the quality of life | at baseline, immediately after treatment completion, 3 and 12 months after treatment completion
  Comparison of the WHOQOL-BREF questionnaire mean between baseline, immediately after treatment the end of the protocol treatment, 3 and 12 months after the end of the protocol treatment. Quantitative evaluation of the primary outcome.
Change in the range of motion | at baseline, immediately after treatment completion, 3 and 12 months after treatment completion
  Comparison of the range of motion between baseline, immediately after the end of the protocol treatment, 3 and 12 months after the end of the protocol treatment. Quantitative evaluation of the primary outcome.
Change in the pressure pain | at baseline, immediately after treatment completion, 3 and 12 months after treatment completion
  Comparison of the pressure pain (algometer) between baseline, immediately after the end of the protocol treatment, 3 and 12 months after the end of the protocol treatment. Quantitative evaluation of the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Justyna Wyszyńska, PhD, Principal Investigator — University of Rzeszow
Locations (1):
- University of Rzeszów, Rzeszów, Poland

IPD SHARING:
Plan to Share IPD: No